CLINICAL TRIAL: NCT05443412
Title: Artificial Intelligence (AI)-Assisted Risk-based Prostate Cancer Detection: A Synergy of Novel Biomarkers, Advanced Imaging, and Robotic-assisted Diagnosis
Brief Title: Artificial Intelligence (AI)-Assisted Risk-based Prostate Cancer Detection
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHIU Ka Fung Peter, Associate Professor, Chinese University of Hong Kong
Other Study IDs: CRE 2022.245
Record Dates: First submitted 2022-06-22; First posted 2022-07-05 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic test for prostate cancer — All recruited patients will undergo investigations including urine for spermine, blood for miRNA, TRUS, and MRI prostate. Patients with high suspicion of Clinically significant prostate cancer in any one step (urine, blood, ultrasound, OR MRI) will be offered an image-guided prostate biopsy.

SUMMARY:
This is a prospective clinical study recruiting 510 men at risk of PCa to undergo urine, blood, AI-assisted ultrasound and AI-assisted MRI investigations to stratify risk of clinically significant PCa (csPCa). (sample size calculation in section 5)

DETAILED DESCRIPTION:
All recruited patients will undergo investigations including urine for spermine, blood for miRNA, TRUS, and MRI prostate. Patients with high suspicion of csPCa in any one step (urine, blood, ultrasound, OR MRI) will be offered an image-guided prostate biopsy. This will be followed by machine learning techniques to find the best combination in predicting csPCa.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥18 years of age
* Clinical suspicion of prostate cancer
* Serum Prostate-specific antigen (PSA) 4-20 ng/mL
* Digital rectal examination ≤ cT2 (organ confined cancer)
* Able to provide written informed consent

Exclusion Criteria:

* Prior prostate biopsy
* Past or current history of prostate cancer
* Contraindicated to undergo plain MRI scan (e.g. pacemaker in-situ, claustrophobia)
* Contraindicated to transperineal prostate biopsy: active urinary tract infection, fail TRUS probe insertion or lithotomy position, uncorrectable coagulopathy, antiplatelet or anticoagulant which cannot be stopped

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All consecutive men referred for elevated PSA 4-20 ng/mL
Sampling Method: Non-Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of clinically significant Prostate cancer (csPCa); • csPCa is diagnosis of ISUP Grade group ≥2 prostate cancer in at least 1 biopsy core | Through study completion, an average of 1 year
  Assessed by by machine learning algorithms utilizing clinical parameters, novel biomarkers and AI-assisted imaging

SECONDARY OUTCOMES:
Diagnosis of any grade of prostate cancer | Through study completion, an average of 1 year
  Assessed by prostate biopsy
Proportion of men with diagnosis of clinically insignificant prostate cancer | Through study completion, an average of 1 year
  Assessed by prostate biopsy
Prostate biopsies that can be avoided | Through study completion, an average of 1 year
  Assessed by using different machine learning algorithms
The concordance of AI-assisted TRUS & MRI diagnosis and biopsy outcomes | Through study completion, an average of 1 year
  Assessed by using different machine learning algorithms and prostate biopsy result

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ka-Fung CHIU, FRCS, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rawla P. Epidemiology of Prostate Cancer. World J Oncol. 2019 Apr;10(2):63-89. doi: 10.14740/wjon1191. Epub 2019 Apr 20. PMID 31068988
- [Background] Hugosson J, Roobol MJ, Mansson M, Tammela TLJ, Zappa M, Nelen V, Kwiatkowski M, Lujan M, Carlsson SV, Talala KM, Lilja H, Denis LJ, Recker F, Paez A, Puliti D, Villers A, Rebillard X, Kilpelainen TP, Stenman UH, Godtman RA, Stinesen Kollberg K, Moss SM, Kujala P, Taari K, Huber A, van der Kwast T, Heijnsdijk EA, Bangma C, De Koning HJ, Schroder FH, Auvinen A; ERSPC investigators. A 16-yr Follow-up of the European Randomized study of Screening for Prostate Cancer. Eur Urol. 2019 Jul;76(1):43-51. doi: 10.1016/j.eururo.2019.02.009. Epub 2019 Feb 26. PMID 30824296
- [Background] Chiu PK, Teoh JY, Chan SY, Chu PS, Man CW, Hou SM, Ng CF. Role of PSA density in diagnosis of prostate cancer in obese men. Int Urol Nephrol. 2014 Dec;46(12):2251-4. doi: 10.1007/s11255-014-0826-7. Epub 2014 Sep 9. PMID 25201460
- [Background] Chiu PK, Roobol MJ, Nieboer D, Teoh JY, Yuen SK, Hou SM, Yiu MK, Ng CF. Adaptation and external validation of the European randomised study of screening for prostate cancer risk calculator for the Chinese population. Prostate Cancer Prostatic Dis. 2017 Mar;20(1):99-104. doi: 10.1038/pcan.2016.57. Epub 2016 Nov 29. PMID 27897172
- [Background] Chiu PK, Ng CF, Semjonow A, Zhu Y, Vincendeau S, Houlgatte A, Lazzeri M, Guazzoni G, Stephan C, Haese A, Bruijne I, Teoh JY, Leung CH, Casale P, Chiang CH, Tan LG, Chiong E, Huang CY, Wu HC, Nieboer D, Ye DW, Bangma CH, Roobol MJ. A Multicentre Evaluation of the Role of the Prostate Health Index (PHI) in Regions with Differing Prevalence of Prostate Cancer: Adjustment of PHI Reference Ranges is Needed for European and Asian Settings. Eur Urol. 2019 Apr;75(4):558-561. doi: 10.1016/j.eururo.2018.10.047. Epub 2018 Nov 2. PMID 30396635
- [Background] Chiu PK, Roobol MJ, Teoh JY, Lee WM, Yip SY, Hou SM, Bangma CH, Ng CF. Prostate health index (PHI) and prostate-specific antigen (PSA) predictive models for prostate cancer in the Chinese population and the role of digital rectal examination-estimated prostate volume. Int Urol Nephrol. 2016 Oct;48(10):1631-7. doi: 10.1007/s11255-016-1350-8. Epub 2016 Jun 27. PMID 27349564
- [Background] Chiu PK, Teoh JY, Lee WM, Yee CH, Chan ES, Hou SM, Ng CF. Extended use of Prostate Health Index and percentage of [-2]pro-prostate-specific antigen in Chinese men with prostate specific antigen 10-20 ng/mL and normal digital rectal examination. Investig Clin Urol. 2016 Sep;57(5):336-42. doi: 10.4111/icu.2016.57.5.336. Epub 2016 Aug 31. PMID 27617315
- [Background] Ng CF, Chiu PK, Lam NY, Lam HC, Lee KW, Hou SS. The Prostate Health Index in predicting initial prostate biopsy outcomes in Asian men with prostate-specific antigen levels of 4-10 ng/mL. Int Urol Nephrol. 2014 Apr;46(4):711-7. doi: 10.1007/s11255-013-0582-0. Epub 2013 Oct 18. PMID 24136184
- [Background] Ng CF, Yeung R, Chiu PK, Lam NY, Chow J, Chan B. The role of urine prostate cancer antigen 3 mRNA levels in the diagnosis of prostate cancer among Hong Kong Chinese patients. Hong Kong Med J. 2012 Dec;18(6):459-65. PMID 23223645
- [Background] de la Taille A, Irani J, Graefen M, Chun F, de Reijke T, Kil P, Gontero P, Mottaz A, Haese A. Clinical evaluation of the PCA3 assay in guiding initial biopsy decisions. J Urol. 2011 Jun;185(6):2119-25. doi: 10.1016/j.juro.2011.01.075. Epub 2011 Apr 15. PMID 21496856
- [Background] Van Neste L, Hendriks RJ, Dijkstra S, Trooskens G, Cornel EB, Jannink SA, de Jong H, Hessels D, Smit FP, Melchers WJ, Leyten GH, de Reijke TM, Vergunst H, Kil P, Knipscheer BC, Hulsbergen-van de Kaa CA, Mulders PF, van Oort IM, Van Criekinge W, Schalken JA. Detection of High-grade Prostate Cancer Using a Urinary Molecular Biomarker-Based Risk Score. Eur Urol. 2016 Nov;70(5):740-748. doi: 10.1016/j.eururo.2016.04.012. Epub 2016 Apr 20. PMID 27108162
- [Background] Desai MM, Cacciamani GE, Gill K, Zhang J, Liu L, Abreu A, Gill IS. Trends in Incidence of Metastatic Prostate Cancer in the US. JAMA Netw Open. 2022 Mar 1;5(3):e222246. doi: 10.1001/jamanetworkopen.2022.2246. PMID 35285916
- [Background] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975
- [Background] Mottet N, van den Bergh RCN, Briers E, Van den Broeck T, Cumberbatch MG, De Santis M, Fanti S, Fossati N, Gandaglia G, Gillessen S, Grivas N, Grummet J, Henry AM, van der Kwast TH, Lam TB, Lardas M, Liew M, Mason MD, Moris L, Oprea-Lager DE, van der Poel HG, Rouviere O, Schoots IG, Tilki D, Wiegel T, Willemse PM, Cornford P. EAU-EANM-ESTRO-ESUR-SIOG Guidelines on Prostate Cancer-2020 Update. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2021 Feb;79(2):243-262. doi: 10.1016/j.eururo.2020.09.042. Epub 2020 Nov 7. PMID 33172724
- [Background] Tsoi TH, Chan CF, Chan WL, Chiu KF, Wong WT, Ng CF, Wong KL. Urinary Polyamines: A Pilot Study on Their Roles as Prostate Cancer Detection Biomarkers. PLoS One. 2016 Sep 6;11(9):e0162217. doi: 10.1371/journal.pone.0162217. eCollection 2016. PMID 27598335
- [Background] Chiu PK, Fung YH, Teoh JY, Chan CH, Lo KL, Li KM, Tse RT, Leung CH, Wong YP, Roobol MJ, Wong KL, Ng CF. Urine spermine and multivariable Spermine Risk Score predict high-grade prostate cancer. Prostate Cancer Prostatic Dis. 2021 Jun;24(2):542-548. doi: 10.1038/s41391-020-00312-1. Epub 2021 Jan 6. PMID 33408349
- [Background] Tsoi TH, Gu YJ, Lo WS, Wong WT, Wong WT, Ng CF, Lee CS, Wong KL. Study of the Aggregation of DNA-Capped Gold Nanoparticles: A Smart and Flexible Aptasensor for Spermine Sensing. Chempluschem. 2017 May;82(5):802-809. doi: 10.1002/cplu.201700155. PMID 31961525
- [Background] Liu HP, Lai HM, Guo Z. Prostate cancer early diagnosis: circulating microRNA pairs potentially beyond single microRNAs upon 1231 serum samples. Brief Bioinform. 2021 May 20;22(3):bbaa111. doi: 10.1093/bib/bbaa111. PMID 32607548
- [Background] Urabe F, Matsuzaki J, Yamamoto Y, Kimura T, Hara T, Ichikawa M, Takizawa S, Aoki Y, Niida S, Sakamoto H, Kato K, Egawa S, Fujimoto H, Ochiya T. Large-scale Circulating microRNA Profiling for the Liquid Biopsy of Prostate Cancer. Clin Cancer Res. 2019 May 15;25(10):3016-3025. doi: 10.1158/1078-0432.CCR-18-2849. Epub 2019 Feb 26. PMID 30808771
- [Background] Grey ADR, Scott R, Shah B, Acher P, Liyanage S, Pavlou M, Omar R, Chinegwundoh F, Patki P, Shah TT, Hamid S, Ghei M, Gilbert K, Campbell D, Brew-Graves C, Arumainayagam N, Chapman A, McLeavy L, Karatziou A, Alsaadi Z, Collins T, Freeman A, Eldred-Evans D, Bertoncelli-Tanaka M, Tam H, Ramachandran N, Madaan S, Winkler M, Arya M, Emberton M, Ahmed HU. Multiparametric ultrasound versus multiparametric MRI to diagnose prostate cancer (CADMUS): a prospective, multicentre, paired-cohort, confirmatory study. Lancet Oncol. 2022 Mar;23(3):428-438. doi: 10.1016/S1470-2045(22)00016-X. PMID 35240084
- [Background] Liu Q, Dou Q, Yu L, Heng PA. MS-Net: Multi-Site Network for Improving Prostate Segmentation With Heterogeneous MRI Data. IEEE Trans Med Imaging. 2020 Sep;39(9):2713-2724. doi: 10.1109/TMI.2020.2974574. Epub 2020 Feb 17. PMID 32078543
- [Background] Chiu PK, Shen X, Wang G, Ho CL, Leung CH, Ng CF, Choi KS, Teoh JY. Enhancement of prostate cancer diagnosis by machine learning techniques: an algorithm development and validation study. Prostate Cancer Prostatic Dis. 2022 Apr;25(4):672-676. doi: 10.1038/s41391-021-00429-x. Epub 2021 Jul 15. PMID 34267331
- [Background] Wery M. [Malaria. Biologic diagnosis. Present status and the future]. Rev Prat. 1988 Jun 16;38(18):1159-63. No abstract available. French. PMID 3051299
- [Background] Shen X, Wang G, Kwan RY, Choi KS. Using Dual Neural Network Architecture to Detect the Risk of Dementia With Community Health Data: Algorithm Development and Validation Study. JMIR Med Inform. 2020 Aug 31;8(8):e19870. doi: 10.2196/19870. PMID 32865498